## Final In-Person Informed Consent Form

Native-Changing High-risk Alcohol Use and Increasing Contraception Effectiveness Study

NCT03930342

Document Date: 9/12/2023

# WASHINGTON STATE UNIVERSITY Research Study Consent Form

**Study Title:** Randomized Trial of an Intervention for Preventing Alcohol-Exposed

Pregnancy among Women in a Remote Reservation Community

#### Researchers:

| Researcher | Title | Affiliation | Phone Number |
|---|---|---|---|
| Dedra Buchwald, MD | Professor<br>and<br>Director | Washington State University, Elson<br>Floyd College of Medicine, Initiative<br>for Research and Education to<br>Advance Community Health | (206) 708-8665 |
| Karen Little Wounded | Research<br>Coordinator | Missouri Breaks Industries<br>Research Inc., Eagle Butte, SD | (605) 964-1260 |
| Marcia O'Leary, RN | Co-<br>Investigator<br>and<br>Manager | Missouri Breaks Industries<br>Research Inc., Eagle Butte, SD | (605) 964-3418 |

**Sponsor:** National Institute on Alcohol Abuse and Alcoholism

You are being asked to take part in a research study. This form tells you about the research study and what will happen if you decide to take part. Please take as much time as you need to read the form carefully. Ask the study staff or researcher to explain anything you don't understand. You can decide not to join the study. If you join the study, you can change your mind later or quit at any time during the study. If you decide not to take part in the study or quit during the study, you will not incur any penalties or loss of services. This study has been approved by the Washington State University Institutional Review Board, the Great Plains Institutional Review Board, and the Cheyenne River Sioux Tribe.

#### What is this study about?

This research study is being done to find out if a program called Native-CHOICES can reduce the risk of alcohol-exposed pregnancies among American Indian women. Native-CHOICES encourages women to reduce their alcohol consumption and use birth control methods. Both of these approaches can reduce alcohol-exposed pregnancies.

You are being asked to take part because you are an American Indian woman living on or near the Cheyenne River Sioux Indian reservation and are between the ages of 18 to 44 years old.

We will ask you some questions to determine if you are eligible. You **cannot** take part in this study if you are:

- Under 18 years old
- Pregnant
- Effectively using birth control
- Unable to get pregnant
- Not using alcohol
- Not sexually active with a male partner
- Living with another person who is already taking part in this study.

## What will I be asked to do if I am in this study?

If you are eligible, you will be randomly selected to receive either Native-CHOICES or be in a control group. The control group will be offered the same Native-CHOICES program after the main part of the study ends. Regardless of whether you receive Native-CHOICES now or later, you should receive usual health care.

Everyone who takes part in the study will be asked to complete a survey at the beginning of the study and 6 weeks, 3 months, and 6 months after you start the study. The survey takes 60 to 90 minutes. You will be asked about your:

- Use of alcohol and tobacco
- Use of birth control
- Health including feelings and relationships
- Background including, age, income, and employment

You do not have to answer any questions that you do not want to answer.

#### Native-CHOICES Group

Women in this group will be asked to:

- Attend 2 Native-CHOICES sessions, each of which is about 90 minutes. In the session, you will meet with a Native-CHOICES coordinator to set goals for yourself and work on the study workbook. You will talk about your alcohol use and birth control goals.
- The sessions may be audio recorded for quality improvement purposes. Your name and identity will not be attached to the recording. The recording will only be used by the research team to make sure the study is being done as planned. Youcan choose to not have your session recorded.
- Attend one visit with a health care provider if you want to discuss birth control
  options. It is up to you whether or not you meet with the provider. This visit may take
  up to 30 minutes of your time.
- Decide whether or not to get text or email messages 1 to 2 times a week for 3 months. These texts would be reminders of your appointments or supportive messages about the goals you set for yourself in the sessions.

### **Control Group**

If you are selected to be in the control group, you will have the option to take part in Native-CHOICES after your study activities are complete.

### Are there any benefits to me if I am in this study?

There may be no direct benefit to you for taking part in the study. Study results may help others in the future.

The study will provide a list of local counseling or other health resources. However, any additional services that you decide to get will be at your own expense.

### Are there any risks to me if I am in this study?

You may experience emotional upset when talking about things like your alcohol consumption, feelings, relationships, and use of birth control.

When we contact you to fill out the 6-week and 3-month survey, we will ask you to find a private space where you can answer questions. If you are not able to find a private space, we will find another time to call. If you are not in a private space, others may be able to hear your answers to the survey.

If you are in Native-CHOICES, you can choose to get text or email messages about your alcohol use and birth control. If other people see your phone or email, they may be able to see these messages.

Other study participants may find out you are in the study if you complete the study procedures at our study offices. We will try to schedule the visits in a way that lowers the chance of other participants seeing you and knowing you are in the study.

The study staff must report any threat you make to seriously harm yourself or someone else. They must also report any suspicion of child abuse or neglect or elder abuse or neglect. If you report a threat to seriously harm yourself or to someone else, or if there isany suspicion of child or elder abuse or neglect, the study staff will be required to report that information to the appropriate authorities.

Study staff are also mandatory reporters following CRST Tribal Ordinance 48. Studystaff are obligated to report any participants who are both pregnant and acutely intoxicated at the time of their visit to local authorities.

The researchers and study staff will do everything possible to protect your information. However, there is a very low chance that study information could be released accidentally.If your study information became known, you could experience negative consequences.

#### Will my information be kept private?

The data for this study will be kept private to the extent allowed by federal and state law. No published results will identify you by name or in any other way.

Under certain circumstances, we may be required to release information that identifies you for internal and external reviews of this project.

Your information, including answers to the survey questions, will be kept separately fromyour name. Procedures are in place to protect your privacy during the study. You will meetin a private room for the Native-CHOICES sessions. The survey you complete will include a study ID and will not include your name. All surveys will be kept in a locked file cabinet,in a locked office, to which only study staff have access. Any electronically stored information will be kept in secure locations. Your study visits will be scheduled to avoid contact with other study participants.

Individuals or groups who will have access to study data include all researchers and studystaff, any committees that the review research, funders of the research (the National Institutes of Health), Missouri Breaks Research Institute Inc., and Washington State University.

To help us protect your information, this study has a Certificate of Confidentiality from the National Institutes of Health. This Certificate guarantees that the research team cannot be forced to provide your name or any identifiable research data or specimens in any Federal or state proceedings unless you agree that we can share it. However, we still must report information to local authorities if we learn about child or elder abuse or neglect, or intent to seriously harm yourself or others. We may also need to respond to requests for information from the Department of Health and Human Services or other federal agencies used for audits or program evaluations.

A description of this clinical trial and a summary of the results will be available online at http://www.clinicaltrials.gov, as required by US law. This website will not include information that can identify you. You can search this website at any time.

The results of this study may be published or presented at professional meetings, but the identities of all research participants will remain anonymous.

The data for this study will be kept for at least 6 years after the end of the study.

## Are there any costs or payments for being in this study?

There will be no costs to you for taking part in this study.

As shown here, you will receive up to \$100 for taking part in this study. You will only receive checks for the activities you finish. If you receive payment, you may be asked to provide your home address.

| Study Activity | Check Amount |
|--------------------|--------------|
| Baseline interview | \$30 |
| 6-week interview | \$20 |

| Total | \$100 |
|-------------------|-------|
| 6-month interview | \$30 |
| 3-month interview | \$20 |

Optional: After enrollment, if you choose to refer someone else to the Native- CHOICES study and that person successfully enrolls in the study, you may be eligible for an additional \$20 check.

The optional components of this study are not essential to your participation in this research. You may choose to participate but if you decline there will be no penalty or loss of services or benefits.

## Who can I talk to if I have questions?

If you have questions about this study or the information in this form, please contactthe Research Coordinator, Karen Little Wounded, Missouri Breaks Industries Research Inc., Eagle Butte, SD (605) 964-1260 or at <a href="mailto:karen.littlewounded@mbiri.com">karen.littlewounded@mbiri.com</a>

You can also contact GPIRB Dewey Ertz, EdD at (605) 341-8647 or toll free at (866)331-5794

You can also contact the researcher – Dr. Dedra Buchwald at Washington State University, Elson S. Floyd College of Medicine, Initiative for Research and Education to Advance Community Health, 1100 Olive Way, Suite 1200, Seattle, WA 98101 or at (20) 708-8622 or at <a href="mailto:dedra.buchwald@wsu.edu">dedra.buchwald@wsu.edu</a>.

If you have questions about your rights as a research participant or would like to report a concern or complaint about this study, please contact the Washington State University Institutional Review Board by phone at (509) 335-7646, or by email at <a href="mailto:irb@wsu.edu">irb@wsu.edu</a>. You may also send sent a letter to Neil 427, PO Box 643143, Pullman, WA 99164-3143.

### What are my rights as a research study volunteer?

Your participation in this research study is completely voluntary. You may choose not to be a part of this study or stop taking part at any time. There will be no penalty to you if you choose not to take part. You may choose not to answer any questions that you do not want to answer.

# What does my signature on this consent form mean?

Your signature on this form means that you:

- Understand the information in this form
- Have had all your questions and concerns addressed by study staff or researchers
- Understand the research study and the potential benefits and risks involved

| Statement of Consent | |
|---|---|
| I give my voluntary consent to take part in this st consent form for my records. | udy. I will be given a copy of this |
| Signature of Participant | Date |
| Printed Name of Participant | |
| Statement of Person Obtaining Informed Con | sent |
| I have carefully explained to the woman taking pocertify that when she signs this form, to the best purpose, procedures, potential benefits, and potential | of my knowledge, she understands the |
| I also certify that she: Speaks the language used to explain this re | |
| <ul> <li>Reads well enough to understand this form and understand when the form is read to he</li> <li>Does not appear to have any problems tha it means to take part in this research.</li> </ul> | er . |
| Signature of Person Obtaining Consent | Date |
| Printed Name of Person Obtaining Consent | Role in the Research Study |